CLINICAL TRIAL: NCT06819644
Title: Optimisation of High Flow Oxygen Therapy Settings During Hypoxaemic Respiratory Distress Based on Non-contact Measurement of Lung Volumes by Depth Camera
Acronym: DiStok
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29BRC22.0105; 2022-A01149-34 (Other: ANSM)
Record Dates: First submitted 2025-01-16; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Hypoxemic Respiratory Failure
Keywords: flow oxygen; lung volume; depth camera
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The control arm will consist of patients with hypoxemic respiratory distress treated by high flow oxygen therapy according to standard procedures.
- interventional (Experimental): The interventional arm will consist of patients with hypoxemic respiratory distress treted by high flow oxygen therapy with adjustement of ventilatory parametres based on lung volume measurements.
  Interventions: Drug: high flow oxygen therapy rate adjusted of lung volumes measured

INTERVENTIONS:
Drug: high flow oxygen therapy rate adjusted of lung volumes measured — Use of a technique based on non-contact measurement of lung volumes by depth camera in order to optimise the use of hihg flow oxygen therapy, with adaptation of the flow rate.
  Arms: interventional

SUMMARY:
The goal of this clinical trial is to validate the interest of a strategy adjusting the flow rate delivered under high-flow oxygen (HFO) therapy according to the lung volumes measured by a new technique, in intensive care patients with hypoxemic respiratory distress (HRD).

The main question it aims to answer is:

"The use of a technique of measurement of lung pulmonary with adjustement to the flow rate can make it possible to limite intubation in patients with HRD in intensive care?" The participants will be the patients admitted in intensive care for HRD with the need for treatment with HFO.

This participants will be randomized in :

* the arm control: treated by high flow oxygen therapy according to standard procedures.
* or in the experimental arm : treated by high flow oxygen therapy with adjustement of ventilatory parametres based on lung volume measurements, obtained by the depth camera.

DETAILED DESCRIPTION:
High-flow oxygen therapy (HFO) is a common technique for the management of patient with hypoxemic respiratory distress in intensive care.The variations in lung volumes induced by the HFO in patients is unknown in clinical routine, in the absence of the availability of a effective measurement technique.

The investigators research team validated a new non-invasive, non-contact technique for measuring lung volumes using depth camera. Using a stereoscopic camera, the patient's chest and abdomen are recognized by a artificial intelligence algorithms. The structures of interest of the chest and the abdomen are the identified and the variation in depth of these points in space allows both the integration of lung volume through automatic calibration procedures, the measurement of respiratory rate and comparaison of movement symetries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypoxemic respiratory distress define by the following 4 criteria:
* Respiratory rate ≥ 25 breaths per minutes
* A ratio of the partial pressure of arterial oxygen (PaO2) to the FiO2 ≤ 300 mmHg while the patient is breathing oxygen at a flow rate of 10 liters per minutes or more
* A partial pressure of arterial carbon dioxide (PaCO2) not higher than 45 mmHg
* An absence of clinical history of underlying chronic respiratory failure

Exclusion Criteria:

* A do-not-intubate order
* Pregnant or lactating woman
* Cardiogenic pulmonary edema
* Exacerbation of asthma
* Hemodynamic instability with use of vasopressor at significant dose (norepinephrine > 0.5 mg/h)
* A Glasgow Coma Scale of 12 points of less
* Contraindications to non-invasive ventilation
* Urgent need for endotracheal intubation
* High flow oxygen therapy started within 48 hours before inclusion
* Patient under legal protection or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Use of intubation within 28 days of randomization | from patient randomization to day 90
  Collection of the use of intubation (Yes/No) in patients

SECONDARY OUTCOMES:
Evaluation of organ dysfunction | up to 28 days after randomization
  daily SOFA score
Evaluation of respiratory therapy | up to 28 days after randomization
  daily ROX Index
Reduced need for ventilatory techniques | from inclusion to day 28
  Number of days without ventilatory support
Mortality | 90 days after inclusion
  Number of death
Collection of data on clinicians' acceptance of the technique and on ergonomics | from patient inclusion to day 90
  Evaluation of ergonomy by the System Usability Scale (SUS). The SUS is based on a Likert scale that allows the user to respond on a 5-point scale from 1:'Strongly disagree' to 5:'Strongly agree'.
Collection of data on clinicians' acceptance of the technique and on ergonomics | from patient inclusion to day 90
  Evaluation of load task by NASA-TLX index
Assessment of patient comfort under high oxygen flow | up to 28 days after randomization
  EVA scale

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - AP-HP - Hôpital Louis Mourier, Colombes
  - AP-HP - Hôpital Henri Mondor, Créteil
  - CH Morlaix, Morlaix
  - CHR Orléans, Orléans
  - CH Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No